CLINICAL TRIAL: NCT02596750
Title: The Effect of Microneedle Pretreatment on Topical Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 252160
Record Dates: First submitted 2015-10-31; First posted 2015-11-04 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Each subject will serve as his or her own control. The right forearm and the left forearm will be randomized through a binary randomization to determine whether the right arm will receive microneedle treatment or sham microneedle treatment (roller with no microneedles). This randomization is developed through code in Excel that will result in binary result of either the value 0 or 1 for each subject. For those subjects assigned a binary code of 0, the right forearm will receive microneedle treatment and the left forearm will receive sham microneedle treatment. For those subjects assigned a binary code of 1, the left forearm will receive microneedle treatment and the right forearm will receive sham microneedle treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microneedle Pretreatment (Active Comparator): One ventral forearm is randomized to receive pretreatment with microneedle rollers that are 200 micrometers in length (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 4 min, 10 min, and 30 min time points.
  Interventions: Device: Microneedle Roller
- Sham Microneedle Pretreatment (Sham Comparator): One ventral forearm is randomized to receive pretreatment with sham microneedle rollers (flat roller without any microneedles) that are 200 micrometers in length (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 4 min, 10 min, and 30 min time points.
  Interventions: Device: Sham microneedle Roller

INTERVENTIONS:
Device: Microneedle Roller — 200 micrometer length microneedles (MR2 roller, Clinical Resolution Laboratories, Inc.) mounted on a disposable roller
  Arms: Microneedle Pretreatment
Device: Sham microneedle Roller — Flat roller without microneedles
  Arms: Sham Microneedle Pretreatment

SUMMARY:
This study evaluates the role of microneedle pretreatment in the speed at which anesthesia develops after application of topical 4% lidocaine.

DETAILED DESCRIPTION:
This study evaluates whether the time to anesthesia with topical 4% lidocaine can be accelerated with the use of microneedle pretreatment. The study will evaluate the anesthesia as a randomized split-body study where each subject serves as their own control. The study will be performed on the volar forearm. Prior to application of the topical 4% lidocaine, one arm will be exposed to a microneedle pretreatment on a microneedle roller and the other arm will be exposed to sham microneedle treatment that will consist of a flat roller with no microneedles. Then pain will be assessed with the use of a spring loaded needle lancet that will be applied at 2 min, 5 min, 10 min, and 30 minutes after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Allergy to lidocaine
* Smokers

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

REFERENCES:
- [Background] Sivamani RK, Stoeber B, Wu GC, Zhai H, Liepmann D, Maibach H. Clinical microneedle injection of methyl nicotinate: stratum corneum penetration. Skin Res Technol. 2005 May;11(2):152-6. doi: 10.1111/j.1600-0846.2005.00107.x. PMID 15807814
- [Background] Sivamani RK, Liepmann D, Maibach HI. Microneedles and transdermal applications. Expert Opin Drug Deliv. 2007 Jan;4(1):19-25. doi: 10.1517/17425247.4.1.19. PMID 17184159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Measure Analysis Population Description: This study incorporated a split body design. 21 participants were studied, each participant had a different treatment on each of their forearms, 42 forearms or data points overall.
Units Other Than Participants: Forearm
Groups:
- Microneedle Treatment: Microneedle treatments consisted of pre-treatment with 200 micrometer microneedle rollers and then application of topical 4% lidocaine.
- Sham Microneedle: Sham microneedle treatments consisted of pre-treatment with flat microneedle rollers (no needles) and then application of topical 4% lidocaine.
Period: Baseline
Arm/Group | Microneedle Treatment | Sham Microneedle
Started (21 participants total started) | 21; 21 Forearm | 21; 21 Forearm
Completed (21 participants total completed) | 21; 21 Forearm | 21; 21 Forearm
Not Completed | 0; 0 Forearm | 0; 0 Forearm
Period: 2 Minutes
Arm/Group | Microneedle Treatment | Sham Microneedle
Started | 21; 21 Forearm | 21; 21 Forearm
Completed | 21; 21 Forearm | 21; 21 Forearm
Not Completed | 0; 0 Forearm | 0; 0 Forearm
Period: 5 Minutes
Arm/Group | Microneedle Treatment | Sham Microneedle
Started | 21; 21 Forearm | 21; 21 Forearm
Completed | 21; 21 Forearm | 21; 21 Forearm
Not Completed | 0; 0 Forearm | 0; 0 Forearm
Period: 10 Minutes
Arm/Group | Microneedle Treatment | Sham Microneedle
Started | 21; 21 Forearm | 21; 21 Forearm
Completed | 21; 21 Forearm | 21; 21 Forearm
Not Completed | 0; 0 Forearm | 0; 0 Forearm
Period: 30 Minutes
Arm/Group | Microneedle Treatment | Sham Microneedle
Started | 21; 21 Forearm | 21; 21 Forearm
Completed | 21; 21 Forearm | 21; 21 Forearm
Not Completed | 0; 0 Forearm | 0; 0 Forearm

BASELINE CHARACTERISTICS:
Population: This study uses a 'split body design' where each participant is measured twice (per physical arm). The participants will be half of the arms because each participant had a split body design and so 21 participants will lead to 42 treatment sites.
Units Other Than Participants: Forearms
Groups:
- Microneedle Pretreatment: One ventral forearm is randomized to receive pretreatment with microneedle rollers that are 200 micrometers in length (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 5 min, 10 min, and 30 min time points.
  Microneedle Roller: 200-micrometer length microneedles (MR2 roller, Clinical Resolution Laboratories, Inc.) mounted on a disposable roller
  Topical 4% lidocaine
- Sham Microneedle Pretreatment: One ventral forearm is randomized to receive pretreatment with sham microneedle rollers (flat roller without any microneedles) (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 5 min, 10 min, and 30 min time points.
  Sham microneedle Roller: Flat roller without microneedles
  Topical 4% lidocaine
- Total: Total of all reporting groups
Arm/Group | Microneedle Pretreatment | Sham Microneedle Pretreatment | Total
Number analyzed (Participants) | 21 | 21 | 21
Number analyzed (Forearms) | 21 | 21 | 42
Age, Continuous [Mean (Full Range); unit: years] | 29 [19 to 59] | 29 [19 to 59] | 29 [19 to 59]
Sex: Female, Male [Count of Units; unit: Forearms] — Population: 21 participants studied, each participant had a different treatment on each of their forearms, 42 forearms overall.
  Forearms
    Female | 0 | 0 | 0
    Male | 21 | 21 | 42
Region of Enrollment [Number; unit: Participants]
  United States | 21 | 21 | 21

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain
Description: 100 mm Visual Analog Scale pain grading. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Time Frame: 2 min
Population: All participants
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Forearms
Groups:
- Active Comparator: Microneedle Pretreatment 1 Ventral Forearm: One ventral forearm is randomized to receive pretreatment with microneedle rollers that are 200 micrometers in length (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 5 min, 10 min, and 30 min time points
- Sham Comparator: Sham Microneedle Pretreatment: One ventral forearm is randomized to receive pretreatment with sham microneedle rollers (flat roller without any microneedles) (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 5 min, 10 min, and 30 min time points.
Arm/Group | Active Comparator: Microneedle Pretreatment 1 Ventral Forearm | Sham Comparator: Sham Microneedle Pretreatment
Number analyzed (Participants) | 21 | 21
Number analyzed (Forearms) | 21 | 21
Units on a Scale | 7 (2) | 12 (3)

2. Primary Outcome: Visual Analog Scale Pain
Description: as for outcome 1
Time Frame: 5 min
Population: All participants
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Forearm
Groups:
- Active Comparator: Microneedle Pretreatment One Ventral Forear: One ventral forearm is randomized to receive pretreatment with microneedle rollers that are 200 micrometers in length (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 5 min, 10 min, and 30 min time points
Arm/Group | Active Comparator: Microneedle Pretreatment One Ventral Forear | Sham Comparator: Sham Microneedle Pretreatment
Number analyzed (Participants) | 21 | 21
Number analyzed (Forearm) | 21 | 21
Units on a Scale | 11 (2.5) | 15 (4)

3. Primary Outcome: Visual Analog Scale Pain
Description: as for outcome 1
Time Frame: 10 min
Population: All participants
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Forearm
Arm/Group | Active Comparator: Microneedle Pretreatment One Ventral Forear | Sham Comparator: Sham Microneedle Pretreatment
Number analyzed (Participants) | 21 | 21
Number analyzed (Forearm) | 21 | 21
Units on a Scale | 8 (3) | 12.5 (3)

4. Primary Outcome: Visual Analog Scale Pain
Description: as for outcome 1
Time Frame: 30 min
Population: All participants
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Forearm
Arm/Group | Active Comparator: Microneedle Pretreatment One Ventral Forear | Sham Comparator: Sham Microneedle Pretreatment
Number analyzed (Participants) | 21 | 21
Number analyzed (Forearm) | 21 | 21
Units on a Scale | 4 (1.3) | 14.4 (3.8)

ADVERSE EVENTS:
Time Frame: Adverse event was collected during the study period of which was one day.
Groups:
- Microneedle Pretreatment: One ventral forearm is randomized to receive pretreatment with microneedle rollers that are 200 micrometers in length (Clinical Resolution Laboratories, Inc.). Then topical 4% lidocaine is applied and pain in assessed after a pain stimulus at the 2 min, 5 min, 10 min, and 30 min time points.
  Microneedle Roller: 200 micrometer length microneedles (MR2 roller, Clinical Resolution Laboratories, Inc.) mounted on a disposable roller
  Topical 4% lidocaine
Arm/Group | Microneedle Pretreatment | Sham Microneedle Pretreatment
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No